CLINICAL TRIAL: NCT04698707
Title: The Role of Supermicrosurgical Lymphaticovenous Anastomosis for Lower Limb Lymphedema - A Retrospective Cohort Study
Brief Title: Role of Supermicrosurgical LVA for Lower Limb Lymphedema
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202001420B0
Record Dates: First submitted 2021-01-05; First posted 2021-01-07 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Lymphedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- lower limb lymphedema patients: This retrospective cohort study enrolled 131 lower limb lymphedema patients including 10 patients who have received VLNT as their primary lymphedema surgery showing minimal post-VLNT improvement (Group I) and 121 patients without previous lymphatic surgery (Group II).
  Interventions: Other: Vascularized lymph node flap transfer; Other: Patients without prior lymphedema surgery

INTERVENTIONS:
Other: Vascularized lymph node flap transfer — Patients who have received VLNT as their primary treatment but with minimal improvement
Other: Patients without prior lymphedema surgery — Patients without prior lymphedema surgery

SUMMARY:
Vascularized lymph node flap transfer (VLNT) was believed to be the treatment of choice for moderate-to-severe lymphedema. Recent publications have supported the use of supermicrosurgical lymphaticovenous anastomosis (LVA) for treating severe lymphedema. This study hypothesizes whether LVA can be performed on post-VLNT patients seeking further improvement.

ELIGIBILITY:
Inclusion Criteria:

* From November 2014 to January 2019
* Lower limb lymphedema patients

Exclusion Criteria:

* Patients who have had previous LVA, liposuction, or excisional therapy such as the Charles procedure were excluded.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From November 2014 to January 2019, a total of 131 lower limb lymphedema patients were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2020-10-05 (Actual); Study Completion 2020-11-19 (Actual)

PRIMARY OUTCOMES:
Magnetic resonance volumetry | 6 months after LVA
  Magnetic resonance volumetry was used for measuring preoperative and postoperative volume changes at least 6-month after LVA.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan